CLINICAL TRIAL: NCT02352558
Title: A Phase Ib Clinical Study of BBI608 for Adult Patients With Advanced, Refractory Hematologic Malignancies
Brief Title: A Study of BBI608 in Adult Patients With Advanced, Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-103HEME; BBI608-103HEM (Other: Sumitomo Dainippon Pharma Oncology, Inc.)
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Hematologic Malignancy
Keywords: Multiple Myeloma; Lymphoma; Acute Myeloid Leukemia; Myelo-Dysplastic Syndrome; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — napabucasin; Dexamethasone; Bortezomib; Imatinib Mesylate; ibrutinib

ARMS (9):
- Arm 1 (Experimental): Patients with multiple myeloma treated with BBI608
  Interventions: Drug: BBI608
- Arm 2 (Experimental): Patients with lymphoma treated with BBI608
  Interventions: Drug: BBI608
- Arm 3 (Experimental): Patients with acute myeloid leukemia or myelo-dysplastic syndrome treated with BBI608
  Interventions: Drug: BBI608
- Arm 4 (Experimental): Patients with chronic myeloid leukemia treated with BBI608
  Interventions: Drug: BBI608
- Arm 5 (Experimental): Patients with multiple myeloma treated with BBI608 and dexamethasone
  Interventions: Drug: BBI608; Drug: Dexamethasone
- Arm 6 (Experimental): Patients with multiple myeloma treated with BBI608 and bortezomib
  Interventions: Drug: BBI608; Drug: Bortezomib
- Arm 7 (Experimental): Patients with chronic myeloid leukemia treated with BBI608 and imatinib
  Interventions: Drug: BBI608; Drug: Imatinib
- Arm 8 (Experimental): Patients with chronic lymphocytic leukemia treated with BBI608
  Interventions: Drug: BBI608
- Arm 9 (Experimental): Patients with chronic lymphocytic leukemia treated with BBI608 and ibrutinib
  Interventions: Drug: BBI608; Drug: Ibrutinib

INTERVENTIONS:
Drug: BBI608 — Patients will receive BBI608 orally twice daily, with doses separated by approximately 12 hours. The starting dose for all cohorts will be 240 mg twice daily. Subsequently, cohorts at alternate dose-levels (480 mg twice daily) may be enrolled as determined by the criteria for dose-escalation.
  Other Names: Napabucasin; BB608; BBI-608
Drug: Dexamethasone — Dexamethasone will be taken orally at a dose level of 40 mg once weekly, on Days 1, 8, 15, and 22 of each Cycle. Patients over the age of 75 years are allowed to begin dexamethasone at a dose of 20 mg once weekly, on Days 1, 8, 15, and 22 of each Cycle. Dexamethasone should be taken with food or milk, and a minimum of 2 hours should separate a dose of dexamethasone from a dose of BBI608.
  Arms: Arm 5
Drug: Bortezomib — Bortezomib will be administered at 1.3 mg/m2/dose as a 3-5 second bolus intravenous (IV) injection or subcutaneous injection twice weekly for 2 weeks (Day 1, 4, 8, and 11) followed by a 10-day rest period (Day 12-21).
  Other Names: Velcade
  Arms: Arm 6
Drug: Imatinib — Imatinib will be taken orally once daily with a meal and a large glass of water. For patients having difficulty swallowing, imatinib can be dissolved in water or apple juice for intake. The dose of imatinib is 400 mg for CML patients in the chronic phase and 600 mg for CML patients in the accelerated phase or in blast crisis. A minimum of 2 hours should separate a dose of imatinib from a dose of BBI608.
  Other Names: Gleevec
  Arms: Arm 7
Drug: Ibrutinib — Ibrutinib will be taken orally once daily with water. Do not open, break, or chew the capsules. The dose of ibrutinib is 420 mg for patients with normal liver function and is 140 mg for patients with mild liver impairment (Child-Pugh class A). A minimum of 2 hours should separate a dose of ibrutinib from a dose of BBI608.
  Other Names: Imbruvica
  Arms: Arm 9

SUMMARY:
This is a multicenter, open label, Phase 1 dose-escalation study of BBI608 administered to patients with relapsed, refractory hematologic malignancies, including multiple myeloma, lymphoma, and others.

ELIGIBILITY:
Major Inclusion Criteria:

1. Signed written informed consent must be obtained and documented according to the International Conference on Harmonisation (ICH) and be in accordance with local regulatory requirements
2. A histologically confirmed hematologic malignancy that is advanced, relapsed, or refractory to standard, currently available anti-cancer treatment options
3. ≥ 18 years of age
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 at dose escalation phase and of ≤ 2 at dose expansion phase
5. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after their last dose
6. Females of childbearing potential must have a negative serum pregnancy test
7. Aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN). Patients whose disease involves the liver and who have laboratory values of AST ≤ 3.5 ULN, AST ≤ 3.5 ULN, and albumin ≥ 35g/L may be enrolled if agreed upon by the Principal Investigator and Medical Monitor for the Sponsor
8. Total bilirubin < 1.5 x ULN, except for cases in which elevation of total bilirubin is due to elevated levels of unconjugated bilirubin consistent with a diagnosis of Gilbert's Syndrome
9. Life expectancy ≥ 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2018-12-14 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Determination of the safety and tolerability of BBI608 administered as monotherapy and in combination with dexamethasone, bortezomib, imatinib or ibrutinib by assessing dose-limiting toxicities (DLTs) | 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetic profile of BBI608 when administered in monotherapy and in combination with dexamethasone, bortezomib, imatinib or ibrutinib as assessed by maximum plasma concentration and area under the curve | -5min, 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 8, 11, 12 hours on day 1, cycles 1 and 2
Pharmacodynamic activity of BBI608 when administered in monotherapy and in combination with dexamethasone, bortezomib, imatinib or ibrutinib as assessed by biomarker analysis | 20 weeks
  Histopathology and Cancer Stem Cell assays will be performed to provide information of the biomarkers on patient blood samples collected on-study, as well as on (if available) bone marrow, other biopsied patient tumor tissue, and archival samples.
Assessment of the preliminary anti-tumor activity by performing tumor assessments | 20 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Indiana University, Indianapolis, Indiana
  - West Clinic, Germantown, Tennessee
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Cancer Care Centers of South Texas - HOAST, San Antonio, Texas
  - Virginia Cancer Specialists, P.C., Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, PC, Vancouver, Washington